CLINICAL TRIAL: NCT06272474
Title: Reliability of Virtual Reproduction of Mandibular Movement for Assessing Occlusal Interferences and Adjustments of Designed and Milled Cad-cam Zirconia Crowns; a Diagnostic Accuracy Trial
Brief Title: Virtual Reproduction of Mandibular Movement for Assessing Occlusal Interferences and Adjustments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0266-07/2021 - 18/07/2021
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Dental Occlusion
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Intervention Model Description: Single group is receiving the two interventional arms
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buccal interocclusal records (Active Comparator)
  Interventions: Other: CAD-CAM zirconia crowns using buccal interocclusal record.
- Lateral interocclusal records (Experimental)
  Interventions: Other: CAD-CAM zirconia crowns using lateral interocclusal records.

INTERVENTIONS:
Other: CAD-CAM zirconia crowns using buccal interocclusal record. — Virtual occlusal interferences adjustment of CAD-CAM zirconia crowns using buccal interocclusal record.
  First, scanning the buccal interocclusal record for each patient with the two arches in maximum intercuspation position (MIP) will be performed. The IOS will immediately reproduce the occlusal state of the digital casts; this method is called the buccal bite registration method (BBR).
  Arms: Buccal interocclusal records
Other: CAD-CAM zirconia crowns using lateral interocclusal records. — Virtual occlusal interferences adjustment of CAD-CAM zirconia crowns using lateral interocclusal record.
  A second scan will be performed for each patient to record lateral mandibular excursion. Then, three STL files will be exported; maxillary arch, mandibular arch at MIP and lateral mandibular excursion
  Arms: Lateral interocclusal records

SUMMARY:
Computer-aided designs have considered dynamic occlusion with virtual articulator systems. However, the process involved is currently lengthy. The simplified transfer of casts from a mechanical to a virtual articulator has required bulky and expensive instruments. Recently, new methods based on mandibular motion tracking using optical devices have been introduced for integrating individual functional movement into occlusal morphology.

The aim of this study: This study will clinically assess the reliability of the virtual reproduction of mandibular movement for detecting occlusal interferences and adjustments of designed and milled CAD-CAM zirconia crowns using a digital occlusal analyzer.

Materials and methods: Intraoral optical impression will be made for thirteen selected patients with endodontically treated maxillary first premolars after abutment preparation followed by buccal and lateral interocclusal records taking. Two zirconia crowns will be fabricated for each patient following regular digital workflow with twenty six zirconia crowns, which will be allocated according to the virtual method of adjustment of occlusal interferences into two groups (Group I: Virtual occlusal interferences adjustment of CAD-CAM zirconia crowns using buccal interocclusal record (n=13) and Group II: Virtual occlusal interferences adjustment of CAD-CAM zirconia crowns using buccal and lateral interocclusal records (n=13)). Then milling and sintering of all crowns will be performed following the manufacturer's instructions. The occlusion of all crowns will be analyzed using an electronic pressure analyzer. All data will be statistically analyzed and discussed in light of the results obtained.

ELIGIBILITY:
Inclusion Criteria:

The patient presented with successful endodontically treated maxillary 1st premolar.

* Patients having class I occlusion.
* Good oral hygiene with no signs of periapical pathology or periodontal disease(24).
* Patient having natural teeth as opposed to dentition.

Exclusion Criteria:

* Pregnancy, which prevents the use of diagnostic x-rays.
* Parafunctional habits.
* Mobility in the abutment teeth more than grade 1.
* Patient presenting allergy to materials being used.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-09-11 (Actual); Primary Completion 2023-12-09 (Actual); Study Completion 2023-12-09 (Actual)

PRIMARY OUTCOMES:
Static occlusal interference | Through study completion, average 12 months
  it is measured at patient's maximum intercuspation using occlusense device
Dynamic occlusal interference | Through study completion, average 12 months
  it is measured at patient's lateral mandibular movement using occlusense device

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt